

### TRIAL STATISTICAL ANALYSIS PLAN

c26500341-01

| BI Trial No.: | 1400-0001 |
|---|---|
| Title: | Safety, tolerability, pharmacokinetics and pharmacodynamics of single rising subcutaneous doses of BI 473494 in healthy male subjects (single-blind, partially randomised, placebo-controlled parallel group design) |
| | Including Protocol Amendment 1 [c11760893-02] |
| Investigational Product: | BI 473494 |
| Responsible trial statisticians: | Phone: Fax: Phone: Fax: |
| Date of statistical analysis plan: | 29 JAN 2019 SIGNED |
| Version: | Final |

**Proprietary confidential information** 

© 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

TSAP for BI Trial No: 1400-0001 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| 1 | , | ΓΔ | RI | $\mathbf{F}$ | OF · | CO | N | NT | rs |
|---|---|----|----|--------------|--------------|----|---|------|----|
| | • | | | 1 1 | <b>\ / </b> | | | <br> | |

| TITLE | PAGE | 1 |
|------------|------------------------------------------------|----|
| 1. | TABLE OF CONTENTS | 2 |
| LIST O | F TABLES | 4 |
| 2. | LIST OF ABBREVIATIONS | 5 |
| 3. | INTRODUCTION | 8 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | 9 |
| 5. | ENDPOINTS | 10 |
| 5.1 | PRIMARY ENDPOINT | 10 |
| 5.2 | SECONDARY ENDPOINTS | |
| 5.2.1 | Key secondary endpoints | |
| 5.2.2 | Secondary endpoints | |
| 6. | GENERAL ANALYSIS DEFINITIONS | 13 |
| 6.1 | TREATMENTS | |
| 6.2 | IMPORTANT PROTOCOL DEVIATIONS | 15 |
| 6.3 | SUBJECT SETS ANALYSED | |
| 6.5 | POOLING OF CENTRES | 18 |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | 19 |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS | |
| 7. | PLANNED ANALYSIS | 22 |
| 7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION | 23 |
| 7.3 | TREATMENT COMPLIANCE | 24 |
| 7.4 | PRIMARY ENDPOINTS | 24 |
| 7.5 | SECONDARY ENDPOINTS | 24 |
| 7.5.1 | Key secondary endpoints | 24 |
| 7.5.2 | Secondary endnoints | 24 |
| 7.7 | EXTENT OF EXPOSURE | 26 |
| <b>7.8</b> | SAFETY ANALYSIS | 26 |
| 7.8.1 | Adverse events | 26 |
| 7.8.2 | Laboratory data | 28 |
| 7.8.3 | Vital signs | 28 |
| 7.8.4 | ECG | 28 |
| 7.8.5 | Others | 29 |
| 8 | REFERENCES | 30 |

| Boehringer Ingelheim |
|---------------------------------|
| TCAD for DI Trial No. 1400 0001 |

| TSAP to | r BI Trial No: 1400-0001 | |
|---|---|---|
| Proprietary c | onfidential information © 2019 Boehringer Ingelheim International GmbH | or one or more of its affiliated companies |
| 10. | HISTORY TABLE | 33 |
| 10. | IIIST STEET TIEEE | |

TSAP for BI Trial No: 1400-0001 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### LIST OF TABLES

| Table 6.1: 1 | Labels for treatments for use in the CTR | |
|--------------|----------------------------------------------|----|
| Table 6.2: 1 | Important protocol deviations | 16 |
| | Analysis sets for endpoints/data description | |
| | Time schedule of 12-lead ECG recordings | |
| | History table | |

TSAP for BI Trial No: 1400-0001

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 2. LIST OF ABBREVIATIONS

| Term | Definition / description |
|---|---|
| ADA | Anti-drug Antibody |
| ADS | Analysis Dataset |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ALT | Alanine Aminotransferase |
| ANCOVA | Analysis of Covariance |
| ANOVA | Analyis of Variance |
| AST | Aspartate Aminotransferase |
| AUC | Area Under The Concentration-Time Curve |
| $AUC_{0-tz}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point |

BI Boehringer Ingelheim

CARE Clinical Analysis and Reporting Environment

CI Confidence Interval

C<sub>max</sub> Maximum measured concentration of the analyte in plasma

CRF Case report form

CTP Clinical Trial Protocol
CTR Clinical Trial Report

CV Arithmetic Coefficient of Variation

DB Dose Proportionality, Between-Subject Design

DBLM Database Lock Meeting
DILI Drug induced liver injury

ECG Electrocardiogram

EudraCT European Union Drug Regulating Authorities Clinical Trials

TSAP for BI Trial No: 1400-0001 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Term | Definition / description |
|---|---|
| gCV | Geometric Coefficient of Variation |
| gMean | Geometric Mean |
| HR | Heart Rate |
| ICH | International Conference On Harmonisation |
| ISF | Investigators Site File |
| iPD | Important Protocol Deviation |
| LLT | Lower Level Term |
| Max | Maximum |
| MedDRA | Medical Dictionary For Regulatory Activities |
| Min | Minimum |
| N | Number non-missing observations |
| O*C | Oracle Clinical |
| P10 | 10th percentile |
| P90 | 90th percentile |
| PD | Pharmacodynamics |
| PDS | Pharmacodynamic Analysis Set |
| PK | Pharmacokinetics |
| PKS | PK Parameter Analysis Set |
| PR | Pulse Rate |
| PT | Preferred Term |
| Q1 | 1st quartile |
| Q3 | 3rd quartile |
| QRS | Complex of three closely related waves on the ECG (Q, R and S wave) |
| QT | Time between start of the Q-wave and the end of the T-wave on the ECG |
| QTc | QT interval corrected for heart rate using the method of Fridericia (QTcF) or Bazett (QTcB) |
| RAGe | Report Appendix Generator system |
| REP | Residual Effect Period |
| RPM | Report Planning Meeting |
| $\mathrm{SAS}^{\circledR}$ | Statistical Analysis System |

TSAP for BI Trial No: 1400-0001 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Term | Definition / description |
|----------|--------------------------------------------------|
| SD | Standard Deviation |
| SOC | System Organ Class |
| TMCP | Translational Medicine and Clinical Pharmacology |
| TS | Treated Set |
| TSAP | Trial Statistical Analysis Plan |
| ULN | Upper Limit of Normal |
| WHO-DD | World Health Organization Drug Dictionary |
| XPKISTAT | Library of SAS® Macros for PK analysis |

TSAP for BI Trial No: 1400-0001

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 3. INTRODUCTION

As per ICH E9 (1), the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This trial statistical analysis plan (TSAP) assumes familiarity with the Clinical Trial Protocol (CTP), including Protocol Amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomisation.

Study data will be stored in a trial database within the Oracle ClinicalTM (O\*C) system.

Pharmacokinetic (PK) parameters will be calculated using Phoenix WinNonlin<sup>TM</sup> software (version 6.3, Certara USA Inc., Princeton, NJ, USA).

The statistical analyses will be performed within the validated Clinical Analysis and Reporting Environment (CARE), including SAS<sup>TM</sup> (current Version 9.4, by SAS Institute Inc., Cary, NC, USA), and a number of SAS<sup>TM</sup>-based tools (e.g., macros for the analyses of AE data or laboratory data; Report Appendix Generator system (RAGe) for compilation/formatting of the Clinical trial Report (CTR) appendices).

TSAP for BI Trial No: 1400-0001

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

All analyses described in the TSAP are outlined in the CTP. The following changes compared to the protocol will be made:

Dose escalation was stopped after the second dose group (75 µg BI 473494). Therefore, all analyses will be performed for the first and second dose group only.

- As there are only two dose groups available, no dose proportionality analysis will be done. Secondary endpoints (AUC $_{0-tz}$  and C $_{max}$  of BI 473494) will be analysed descriptively only.
- As there are only two dose groups available and only little exposure levels expected, no ECG exposure-repsonse analyses will be done.

As an abbreviated CTR will be written, the change from baseline in body weight will be analysed descriptively only.

### 5. ENDPOINTS

### 5.1 PRIMARY ENDPOINT

**Section 5.2.1 of the CTP:** Primary endpoint to assess safety and tolerability of BI 473494 is the number [N (%)] of subjects with drug-related adverse events.

### 5.2 SECONDARY ENDPOINTS

### 5.2.1 Key secondary endpoints

This section is not applicable as no key secondary endpoints have been defined in the CTP.

### 5.2.2 Secondary endpoints

**Section 5.5.1.1 of the CTP:** *The following pharmacokinetic parameters will be determined for BI 473494 if feasible:* 

- $AUC_{0-tz}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point)
- $C_{max}$  (maximum measured concentration of the analyte in plasma)

TSAP for BI Trial No: 1400-0001 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1400-0001 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENTS

It was planned that in total 88 healthy male subjects participate in the trial, according to 11 sequential groups comprising 8 subjects per group (6 on active drug and 2 on placebo).

For details of dosage and formulation see Table 6.1: 1 below.

Table 6.1: 1 Labels for treatments for use in the CTR

| Trea | Treatment | |
|------|-------------------------------------------|-----------|
| P* | Placebo solution, sc, qd | Placebo |
| A | BI 473494, solution for injection, 35 ug | BI 35 ug |
| В | BI 473494, solution for injection, 75 ug | BI 75 ug |
| C | BI 473494, solution for injection, 150 ug | BI 150 ug |
| D | BI 473494, solution for injection, 300 ug | BI 300 ug |
| E | BI 473494, solution for injection, 550 ug | BI 550 ug |
| F | BI 473494, solution for injection, 1.0 mg | BI 1.0 mg |
| G | BI 473494, solution for injection, 1.6 mg | BI 1.6 mg |
| Н | BI 473494, solution for injection, 2.6 mg | BI 2.6 mg |
| I | BI 473494, solution for injection, 4.0 mg | BI 4.0 mg |
| J | BI 473494, solution for injection, 6.0 mg | BI 6.0 mg |
| K | BI 473494, solution for injection, 8.5 mg | BI 8.5 mg |

<sup>\*:</sup> The placebo control group in the safety evaluation will consist of all placebo treated subjects, regardless of the dose group in which they were treated.

Dose escalation was stopped after the second dose group (Treatment B /  $75\mu g$  BI 473494). Therefore, all analyses will be performed for the first and second dose group only (treatments Placebo,  $35\mu g$  BI 473494 and  $75\mu g$  BI 473494).

The following separate study phases will be defined for the analyses of AEs:

- **Screening** (ranging from 0:00 h on day of informed consent until administration time of study drug (BI 473494 or Placebo))
- On treatment
  - **BI 473494/Placebo treatment** (separately for each treatment, ranging from the time of administration of BI 473494 / Placebo until 0:00h on the day after trial termination date)

Please note that all AEs reported between start of trial drug administration and the last perprotocol contact will be considered on treatment (i.e. no follow-up period is considered in this trial).

Displays of AEs will be presented separately for the treatments Placebo, 35µg BI 473494 and 75µg BI 473494.

Two types of AE displays will be provided in the report:

**A)** Section 15.3 and Appendix 16.1.13.1.8 (for ClinicalTrials.gov and EudraCT only) of the CTR displays:

In these displays, the on treatment phase will be analysed (labelled with the name of the study treatment (short label)). Screening will not be included in this analysis. The following total will be provided in addition (Section 15.3 only):

- a total over all BI 473494 treated phases ("BI Total")
- a total over all on treatment phases included in this analysis ("**Total on treatment**") (Section 15.3 only)
- **B)** Section 15.4 and Appendix 16.1.13.1.8 (except for ClinicalTrials.gov and EudraCT) of the CTR displays:
  - Screening
  - On treatment (labelled with the name of the study treatment (short label))

In Section 16.1.13.1.8 AE tables, the following totals will be provided in addition:

- a total over all BI 473494 treated phases ("BI Total")
- a total over all study phases ("Total")

Tables of vital signs and laboratory values will present results by the above mentioned on treatment phase.

For detailed information on the handling of the treatments in the O\*C views refer to Technical TSAP ADS (analysis data set) plan and Analysis Data Reviewers guide.

#### 6.2 IMPORTANT PROTOCOL DEVIATIONS

Data discrepancies and deviations from the CTP will be identified for all treated subjects.

Consistency check listings (for identification of deviations of time windows) and a list of protocol deviations (e.g. deviations in drug administration, in blood sampling times, etc.) will be provided to be discussed at the Report Planning Meeting and database lock meeting (RPM/DBLM). At this meeting, all manual deviations identified at the sites by the CRAs and deviations too complex to program will be reviewed by the trial team to decide which are considered important. For definition of important protocol deviations (iPD), and for the process of identification of these, refer to the Boehringer Ingelheim (BI) SOP "Identify and Manage Important Protocol Deviations (iPD)" (2).

If any iPDs are identified, they are to be summarised into categories and will be captured in the RPM/DBLM minutes via an accompanying Excel spreadsheet (3). The following Table 6.2.1 contains the categories which are considered to be iPDs in this trial. If the data show other iPDs, this table will be supplemented accordingly by the time of the RPM/DBLM at the latest.

The iPDs will be summarised and listed.

TSAP for BI Trial No: 1400-0001 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Important protocol deviations Table 6.2: 1

| Cat<br>/Cc | tegory<br>ode | Description |
|---|---|---|
| A | | Entrance criteria not met |
| | A1 | Inclusion criteria violated |
| | A2 | Exclusion criteria violated |
| В | | Informed consent |
| | B1 | Informed consent not available |
| | B2 | Informed consent too late |
| C | | Trial medication and randomisation |
| | C1 | Incorrect trial medication taken |
| | C2 | Randomisation not followed |
| | С3 | Non-compliance |
| D | | Concomitant medication |
| | D1 | Concomitant medication with the potential to affect the assessment of the trial medication |
| E | | Missing data |
| | E1 | Certain deviations from procedures used to measure secondary data |
| F | | Incorrect timing <sup>1</sup> |
| | F1 | Certain deviations from time schedule used to measure secondary data |
| G | | Other trial specific important deviations |
| | G1 | Appropriate fasting condition not met prior to study drug administration |
| | G2 | Protocol deviations affecting safety and rights |

Time deviations will only be flagged as iPD, when leading to exclusion of the entire subject from an analysis set

#### 6.3 SUBJECT SETS ANALYSED

TSAP for BI Trial No: 1400-0001

• Treated set (TS):

This subject set includes all subjects who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.

This is the full analysis set population in the sense of ICH-E9 (1).

It is used for demographics, baseline characteristics, and safety analyses.

The ECG analyses are performed on the TS.

**Section 7.3.2 of the CTP:** Pharmacokinetic parameters of a subject will be included in the analysis unless the subject has an important protocol deviation relevant for the evaluation. Whether a protocol deviation is important will be decided no later than in the Report Planning Meeting.

Reasons for exclusion of single pharmacokinetic parameters may be:

- The subject experiences emesis at or before two times median  $t_{max}$ . Median  $t_{max}$  is to be determined for the test product excluding the subjects experiencing emesis.
- The subject experiences emesis at any time during the labelled dosing interval.
- Time deviations
- *Use of restricted medications*

The subject set for the evaluation of PK endpoints [...] will include all treated subjects that provide at least one observation for at least one secondary endpoint without important protocol deviations with respect to the statistical evaluation of PK endpoints.

• PK parameter analysis set (PKS):

The PK parameter analysis set (PKS) includes all subjects from the TS receiving BI 473494 who provide at least one secondary PK parameter that was not excluded according to the description above.

**Section 7.3.2 of the CTP:** *It will be decided in the Report Planning Meeting which subjects are to be included in the PKS.* 

Excluded subjects will be listed with their individual plasma concentrations and individual pharmacokinetic parameters, however, will not be included in descriptive statistics for plasma concentrations, pharmacokinetic parameters or other statistical assessment.

The descriptive analysis of PK concentrations will be based on the analysis data set (ADS) ADPC as described at the beginning of Section 7.

TSAP for BI Trial No: 1400-0001 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 6.3: 1 Analysis sets for endpoints/data description

| Endpoint/data description | | Analysis set | | |
|---|---|---|---|---|
| | | TS | PKS | PDS |
| Primary and further safety endpoints (incl. ECG) | | X | | |
| Secondary | PK endpoints | | X | |
| Demographic/baseline data | | X | | |
| Important protocol deviations | | X | | |
| Disposition | | X | | |

#### 6.5 **POOLING OF CENTRES**

This section is not applicable, because the study was performed in only one centre.

TSAP for BI Trial No: 1400-0001

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

Handling of missing data and outliers will be performed as described in the CTP, Section 7.4.

The only exception where imputation might be necessary for safety evaluation is AE dates. Missing or incomplete AE dates are imputed according to BI standards (see 001-MCG-156 RD-01 (4)).

Missing data and outliers of PK data are handled according to BI standards (see 001-MCS-36-472 RD-01) (5).

If single cardiac cycles of an ECG (out of the generally four) are missing, the arithmetic mean for this single ECG will be computed with the reduced (1, 2 or 3) number of cardiac cycles.

If replicate ECG recordings are missing, the arithmetic means per time point will be computed with the reduced number (1 or 2) of recordings.

For the classification of the on-treatment QTc/QT intervals into "no new onset" / "new onset" categories, a missing value is obtained only in case that

- (i) all on-treatment values are missing and
- (ii) the baseline value is less than or equal to 500 msec, or missing. If condition (i) is fulfilled but the baseline value is greater than 500 msec, this case will be categorized as 'no new onset'. If baseline is missing and the maximum on treatment QTc interval is greater than 450 msec (or 500 msec for QT interval, respectively), this is classified as a 'new onset' in the respective category. If baseline is missing and the maximum QTc interval is less than or equal to 450 msec (or 500 msec for QT interval, respectively), this will be categorized as 'no new onset'. If baseline is missing, a QTc/QT interval > 500 msec at any time on treatment will be a notable finding.

### 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

For vital signs or laboratory measurements, baseline is defined as the last measurement before drug administration (BI or Placebo).

**Section 6.1 of the CTP:** Exact times of measurements outside the permitted time windows will be documented. The acceptable time windows for screening and end of trial examination are given in the CTP Flow Chart.

Study measurements and assessments scheduled to occur 'before' trial medication administration on Day 1 of Visits 2 or 3 are to be performed and completed within a 2 h-period prior to the trial drug administration (including blank values for PK

Starting from 96 h post administration a deviation from the scheduled time for PK sampling ECG and blood sampling for ADA of  $\pm$  70 min is acceptable. However, ECGs should always be time-matched with blood PK sampling.

The acceptable deviation from the scheduled time for vital signs and laboratory tests will be  $\pm 30$  min for the first 72 h after trial drug administration. Starting from 96 h post

administration a deviation from the scheduled time for vital signs and laboratory tests of  $\pm$  70 min is acceptable.

Adherence to time windows will be checked via the consistency check listings at the RPM/DBLM.

There will be a centralised evaluation of the 12-lead ECG recordings at the time points and for the ECG recordings specified in the Table 6.7: 1 below:

Table 6.7: 1 Time schedule of 12-lead ECG recordings

| Visit | Day | Planned time [hh:mm] (relative to drug administration) | Study phase | Central evaluation |
|---|---|---|---|---|
| 1 | -21 to -2 | | Screening | NA |
| 2 | -1 | -24:00 | | NA |
| 3 | 1 | -1:00 | | first of three replicate ECG |
| | | -0:45 | | first of three replicate ECG |
| | | -00:30 | | first of three replicate ECG |
| | | 06:00 | On treatment | first of three replicate ECG |
| | | 09:00 | | first of three replicate ECG |
| | | 12:00 | | first of three replicate ECG |
| | 2 | 24:00 | | first of three replicate ECG |
| | | 28:00 | | first of three replicate ECG |
| | | 34:00 | | first of three replicate ECG |
| | 3 | 48:00 | | first of three replicate ECG |
| | | 60:00 | | first of three replicate ECG |
| | 4 | 72:00 | | first of three replicate ECG |
| | 5 | 96:00 | | first of three replicate ECG |
| | 6 | 120:00 | | first of three replicate ECG |
| | 8 | 168:00 | | first of three replicate ECG |
| | 11 | 240:00 | | first of three replicate ECG |
| | 15 | 336:00 | | first of three replicate ECG |
| | 22 | 504:00 | | first of three replicate ECG |
| | 29 | 672:00 | | first of three replicate ECG |
| 4 | 33 to 40 | | End of trial examination | NA |

Triple ECGs (3 single ECGs of 10 sec duration each, recorded within 180 sec) will be recorded at all time points, except for Screening, planned time -24:00h and End-of-trial visit.

At these time-points single ECGs will be recorded. Three pre-dose triplicate ECGs within 60 minutes are to be recorded as baseline.

**Section 6.1 of the CTP:** Only the first of the three replicate ECGs at a single time point or at baseline will be evaluated.

The baseline value of an ECG variable is defined as the mean of the first single ECG measurement of each triple ECG prior to first drug administration.

#### 7. PLANNED ANALYSIS

The placebo group in the safety evaluation will consist of all placebo treated subjects, regardless of the dose group in which they were treated.

Safety analysis (refer to Section 7.8) will be performed by and will be presented in Sections 15.1 to 15.4 of the CTR and in Appendix 16.2 and 16.1.13.1.

Descriptive data analysis of PK parameters and concentrations will be performed by the department Translational Medicine and Clinical Pharmacology (TMCP) at BI and will be presented in Section 15.6 and 15.7 of the CTR.

The format of the listings and tables will follow the standards defined in the BI corporate guideline "Reporting of Clinical Trials and Project Summaries" [001-MCG-159] (6) with the exception of those generated for PK-calculations.

The individual values of all subjects will be listed, sorted by treatment group, subject number, and visit.

The listings will be included in Appendix 16.2 of the CTR.

For end-of-text tables, the set of summary statistics for non-PK parameters is:

N number non-missing observations

Mean arithmetic mean SD standard deviation

Min minimum Median median Max maximum

For analyte concentrations, the following descriptive statistics will additionally be calculated:

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

For PK parameters, the following descriptive statistics will additionally be calculated:

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

P10 10th percentile Q1 1st quartile Q3 3rd quartile P90 90th percentile

The data format for descriptive statistics of concentrations will be identical with the data format of the respective concentrations. The descriptive statistics of PK parameters will be calculated using the individual values with the number of decimal places as provided by the evaluation program. Then the individual values as well as the descriptive statistics will be reported with three significant digits in the CTR.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category, as well as the percentage (%) for each treatment group. Percentages will be rounded to one decimal place and will be based on all subjects in the respective subject set whether they have non-missing values or not. The category 'missing' will be displayed only if there are actually missing values.

Units of variables should be given in the titles or column/row descriptors in square brackets (e.g. [mg]).

#### Exclusion of PK parameters

The analysis data set (ADS) ADPP contains column variables APEXC and APEXCO indicating inclusion/exclusion (APEXC) of a PK parameter and an analysis flag comment (APEXCO). All analyses based on the PKS will include parameters if they are not flagged for exclusion, that is APEXCO is equal to "Included".

#### Exclusion of PK concentrations

The ADS ADPC (PK concentrations per time-point or per time-interval) contains column variables ACEXC or ACEXCO indicating inclusion/exclusion (ACEXC) of a concentration and an analysis flag comment (ACEXCO). Exclusion of a concentration depends on the analysis flag comment ACEXCO. For example, if ACEXCO is set to 'ALL CALC', the value will be excluded for all types of analyses based on concentrations. If ACEXCO is set to 'DESC STATS' the value will be excluded from descriptive evaluations per planned time point/ time interval. If ACEXCO contains the addition 'TIME VIOLATION' or 'TIME DEVIATION' the value can be used for further analyses based on actual times. If ACEXCO is set to 'HALF LIFE' the value will be excluded from half-life calculation (and, as a consequence, any calculation that relies on  $\lambda_z$ ) only; the value is included for all other analyses.

Further details are given in 001-MCS-36-472\_RD-01 "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies" (5) and 001-MCS-36-472\_RD-03 "Description of Analytical Transfer Files and PK/PD Data Files" (11).

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the report, based on the TS. The data will be summarized by treatment group and in total.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Frequency tables are planned for this section of the report, based on the TS.

Concomitant diseases will be coded using the coding system of the Medical Dictionary for Drug Regulatory Activities (MedDRA). Medications will be coded using the latest version of the World Health Organization Drug Dictionary (WHO-DD). The coding version number will be displayed as a footnote in the respective output.

The diagnoses and medications will be listed. Subjects without any concomitant diagnoses or concomitant therapies should be marked with a "No" in the respective column.

The relevance of the concomitant therapies to the evaluation of PK will be decided no later than at the RPM/DBLM.

#### 7.3 TREATMENT COMPLIANCE

**Section 4.3 of the CTP:** Compliance will be assured by administration of all trial medication in the study centre under supervision of the investigating physician or a designee. The measured plasma concentrations of investigational and non-investigational medicinal products and urinary excretion of BI 473494 will provide additional confirmation of compliance.

It is not intended to list the compliance separately. Any deviations from complete intake will be addressed in the RPM/DBLM (cf. TSAP <u>Section 6.2</u>) and described in the CTR.

#### 7.4 PRIMARY ENDPOINTS

Refer to TSAP <u>Section 7.8</u> for a description of the analysis of safety and tolerability of BI 473494.

#### 7.5 SECONDARY ENDPOINTS

### 7.5.1 Key secondary endpoints

This section is not applicable as no key secondary endpoint has been specified in the protocol.

### 7.5.2 Secondary endpoints

Descriptive statistics of plasma concentrations and PK endpoints will be done by the department TMCP at BI and will be presented in Section 15.6 of the CTR.

The analysis of PK parameters as well as the tables and graphs for the pharmacokinetic non-compartmental analyses will follow specific definitions of this TSAP or, otherwise, the BI standard procedure "Standards and processes for analyses performed within Clinical Pharmacokinetics/Pharmacodynamics" [001-MCS-36-472] (7).

TSAP for BI Trial No: 1400-0001 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.7 EXTENT OF EXPOSURE

Descriptive statistics are planned for this section of the report based on the TS. The date and time of drug administration will be listed for each subject.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the TS.

If not stated otherwise, the safety results will be sorted by treatment group. The safety data for treated subjects who failed to complete the study (dropouts or withdrawals) will be reported as far as their data are available. All withdrawals will be documented and the reason for withdrawal recorded.

#### 7.8.1 Adverse events

AEs will be coded with the most recent version of MedDRA.

The analyses of AEs will be descriptive in nature and will be based on BI standards as presented in the corporate guideline: "Analysis and Presentation of Adverse Event Data from Clinical Trials" [001-MCG-156] (8).

The standard AE analyses will be based on the number of subjects with AEs (and not on the number of AEs).

For analysis multiple AE occurrence data on the CRF will be collapsed into an AE provided that all of the following applies:

- All AE attributes are identical (LLT, intensity, action taken, therapy required, seriousness, reason for seriousness, relationship, outcome, AE of special interest)
- The occurrences were time-overlapping or time-adjacent (time-adjacency of two occurrences is given if the second occurrence started within one hour after end of the first occurrence).

For further details on summarization of AE data, please refer to [001-MCG-156] (8,4).

**Section 5.2.2.1 of the CTP:** *The following are considered as AESIs in this trial:* 

- <u>Hepatic injury:</u> A hepatic injury is defined by the following alterations of hepatic laboratory parameters:
  - an elevation of AST (aspartate aminotransferase) and/or ALT (alanine aminotransferase) ≥3-fold ULN combined with an elevation of total bilirubin ≥2-fold ULN measured in the same blood sample, and/or

TSAP for BI Trial No: 1400-0001

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

• aminotransferase (ALT, and/or AST) elevations ≥10 fold ULN

These lab findings constitute a hepatic injury alert and the patients showing these lab abnormalities need to be followed up according to the 'DILI checklist' provided in the ISF. In case of clinical symptoms of hepatic injury (icterus, unexplained encephalopathy, unexplained coagulopathy, right upper quadrant abdominal pain, etc.) without lab results (ALT, AST, total bilirubin) available, the Investigator should make sure these parameters are analysed, if necessary in an unscheduled blood test. Should the results meet the criteria of hepatic injury alert, the procedures described in the DILI checklist should be followed.

The analysis of adverse events will be based on the concept of treatment emergent adverse events.

**Section 5.2.2.2 of the CTP:** The REP for BI 473494, when measurable drug levels or PD effects are still likely to be present after the last administration, is not known for this first-in-human trial. Therefore, all AEs reported until the end of trial examination (last per protocol contact) will be considered on treatment [...].

For more details see the TSAP ADS plan.

According to ICH E3 (9), AEs classified as 'other significant' needs to be reported and will include those non-serious and non-significant adverse events with

- (i) 'action taken = discontinuation' or 'action taken = reduced', or
- (ii) marked haematological and other lab abnormalities or lead to significant concomitant therapy as identified by the Clinical Monitor/Investigator at the RPM at the latest.

An overall summary of AEs (including AESIs) will be presented.

The frequency of subjects with AEs will be summarised by treatment, primary system organ class (SOC) and preferred term (PT). Separate tables will be provided for subjects with other significant AEs according to ICH E3 (9), for subjects with serious AEs, for subjects with drug-related AEs, for subjects with drug related serious adverse events and for subjects with AESIs.

The SOC and PTs will be sorted by frequency (within SOC). The MedDRA version number will be displayed as a footnote in the respective output.

In addition, frequencies of subjects with non-serious AEs that had an incidence of > 5% for at least one treatment will be summarised by treatment, primary SOC and PT.

For disclosure of adverse events on EudraCT additional information not included in a standard AE analysis will be performed. The following three entries will be created:

- Adverse Events per arm for disclosure on EudraCT
- Non-serious Adverse Events for disclosure on EudraCT
- Serious Adverse Events for disclosure on EudraCT

#### 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards [001-MCG-157] (10).

Laboratory data will be analysed qualitatively via comparison of laboratory data to their reference ranges. Values outside the reference range as well as values defined as possible clinically significant will be flagged in the data listings.

It is the investigator's responsibility to decide whether a lab value is clinically significant abnormal or not (at the RPM/DBLM at the latest).

#### 7.8.3 Vital signs

Descriptive statistics over time including change from baseline will be performed for vital signs (blood pressure and pulse rate as well as body weight).

#### **7.8.4** ECG

#### 12-lead ECG

Abnormal findings will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator.

All evaluations of ECG data will be based on the TS.

#### Listing of individual data

For all quantitative endpoints, listings of individual data will be shown in Appendix 16.2. For QTcB and RR only listings will be provided. Occurrences of notable findings will be flagged.

Comments regarding the ECGs will be listed.

#### Categorical endpoints

For the categorical endpoints, frequency tables will be provided.

For all subjects with any notable finding in ECG intervals, a separate listing will be created as end-of-text display (based on the same display template as in Appendix 16.2), and the corresponding time profiles will be shown.

#### Quantitative endpoints

Descriptive statistics (N, mean, SD, min, median, max) will be provided for the changes from baseline over time of QTcF, HR, QT, PR and QRS. The time profiles of mean and SD for the changes from baseline on treatment will be displayed graphically by treatment.

#### 7.8.5 **Others**

### Physical examination

Physical examination findings will be reported as relevant medical history/baseline condition (i.e., a condition already existent before intake of study drug) or as AE and will be summarised as such. No separate listing or analysis of physical examination findings will be prepared.

TSAP for BI Trial No: 1400-0001 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **REFERENCES** 8.

| 1. | CPMP/ICH/363/96: "Statistical Principles for Clinical Trials", ICH Guideline Topic E9, |
|---|---|
| | Note For Guidance on Statistical Principles for Clinical Trials, current version. |
| 2. | 001-MCS-40-413: "Identify and Manage Important Protocol Deviations (iPD)", current |
| | version, BIRDS |
| 3. | BI-KMED-COPS-TMP-0001: "iPD log", current version; KMED |
| 4. | 001-MCG-156 RD-01: "Handling of Missing and Incomplete AE Dates", current |
| | version; IDEA for CON. |
| 5. | 001-MCS-36-472_RD-01: "Noncompartmental Pharmacokinetic/Pharmacodynamic |
| | Analyses of Clinical Studies", current version; IDEA for CON. |
| 6. | 001-MCG-159: "Reporting of Clinical Trials and Project Summaries", current version; |
| | IDEA for CON. |
| 7. | 001-MCS-36-472: "Standards and processes for analyses performed within Clinical |
| | Pharmacokinetics/Pharmacodynamics", current version; IDEA for CON. |
| 8. | 001-MCG-156: "Analysis and Presentation of Adverse Event Data from Clinical Trials", |
| | current version; IDEA for CON. |
| 9. | CPMP/ICH/137/95: "Structure and Content of Clinical Study Reports", ICH Guideline |
| | Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current |
| | version. |
| 10. | 001-MCG-157: "Handling, Display and Analysis of Laboratory Data", current version; |
| | IDEA for CON. |
| 11. | 001-MCS-36-472_RD-03: "Description of Analytical Transfer Files and PK/PD Data |
| | Files", current version; IDEA for CON. |
| 12. | Ring A. Statistical models for heart rate correction of the QT interval. Stat Med 2010 |
| | [R10-2920] |

TSAP for BI Trial No: 1400-0001 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1400-0001 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 10. **HISTORY TABLE**

Table 10: 1 History table

| Version | Date | Author | Sections | Brief description of change |
|---|---|---|---|---|
| | (DD-MMM-YY) | | changed | |
| Final | 29-JAN-19 | | None | This is the final TSAP without any |
| | | | | modification |